CLINICAL TRIAL: NCT00524199
Title: The Effects of 12 mg/kg Intravenous Mesna on Plasma Total Homocysteine Concentration in Patients With End-stage Renal Disease Requiring Hemodialysis
Brief Title: Effects of Mesna on Homocysteine in Kidney Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R-06-472; 122006
Record Dates: First submitted 2007-08-30; First posted 2007-09-03 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: End Stage Renal Disease
Keywords: homocysteine; hemodialysis; mesna
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mesna; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline IV infusion over five minutes at the beginning of dialysis.
  Interventions: Other: Saline
- Mesna (Active Comparator): 12 mg/kg mesna IV infusion over five minutes at the beginning of dialysis.
  Interventions: Drug: Mesna

INTERVENTIONS:
Drug: Mesna — 12 mg/kg IV infusion over five minutes at the beginning of dialysis thrice weekly.
  Other Names: Mesnex; Uromitexan
  Arms: Mesna
Other: Saline — Saline IV infusion over five minutes at the beginning of dialysis thrice weekly.
  Arms: Placebo

SUMMARY:
The purpose of this research study is to examine the effect of a drug called mesna on the removal of homocysteine from blood during dialysis. Homocysteine is an amino acid (protein building block) found in the blood of all people, however it is considerably elevated in dialysis patients. People with increased levels of homocysteine in their blood are at increased risk of developing plaque buildup in their arteries and other related problems such as heart attack and stroke. This study will determine if mesna can improve the rate of homocysteine removal from blood during dialysis.

DETAILED DESCRIPTION:
Homocysteine is a thiol amino acid derived from dietary methionine. Elevated plasma total homocysteine (tHcy), termed hyperhomocysteinemia, is a graded, independent risk factor for the development of atherosclerosis. Elevated plasma tHcy can be normalized by supplementation with folic acid and vitamins B6 and B12 in most patients with normal renal function and this treatment has been shown to halt the progression of atherosclerotic plaque.

Over 90% of patients with end-stage renal disease (ESRD) requiring hemodialysis have elevated plasma tHcy. The leading causes of morbidity and mortality in these patients are cardiovascular-related pathologies such as myocardial infarction and stroke. Vitamin supplementation consistently fails to normalize elevated plasma tHcy in patients with ESRD, thus leaving them at increased risk. Plasma tHcy is 70 - 80% covalently protein bound limiting the effectiveness of dialysis as a tHcy lowering treatment.

Mesna (sodium 2-mercaptoethanesulfonic acid) is a thiol-containing drug currently indicated to prevent hemorrhagic cystitis associated with ifosfamide chemotherapy. Mesna has incidentally been shown to deplete plasma thiols in cancer patients undergoing ifosfamide chemotherapy. Mesna acts to exchange with thiols bound to plasma proteins enhancing their renal excretion. In vitro studies in our laboratory have shown that mesna rapidly (within 5 minutes) exchanges with protein bound homocysteine yielding a significantly larger dialyzable fraction of the thiol amino acid.

A pilot study recently completed by our group demonstrated a significant decrease in tHcy in eight hemodialysis patients receiving 12 mg/kg mesna three times a week pre-dialysis for one week. Although this therapy did cause a significant decline in tHcy, mesna failed to reduce tHcy to normal levels. The cumulative effects of mesna administration over a longer treatment period should be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease who have received hemodialysis thrice weekly for at least 90 days
* Serum albumin > 30 g/L.

Exclusion Criteria:

* Patients who refuse to sign a letter of informed consent
* Women who are or are trying to become pregnant or are breast-feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Difference in plasma total homocysteine between placebo and mesna treatments | Four weeks

SECONDARY OUTCOMES:
Excretion of mesna during hemodialysis | duration of dialytic session

CONTACTS AND LOCATIONS:
Overall Officials: David J Freeman, MSc, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's; Andrew A House, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada